CLINICAL TRIAL: NCT03864159
Title: Efficacy of an Intervention Using the Suction Cups and the Foam Roller in the Improvement of the Flexibility of the Ischiotibial Musculature in Basketball Players From 18 to 25 Years Old. A Randomized Clinical Study
Brief Title: Suction Cups and Foam Roller in the Improvement of the Flexibility in Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FLEX
Record Dates: First submitted 2019-03-04; First posted 2019-03-06 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Flexibility, Waxy
Keywords: Cupping therapy; Foam roller; Basketball; Flexibility; Hamstring
MeSH Terms: conditions — Catalepsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suction cups (Experimental): The technique will be performed with the subject sitting on the floor, placing the Foam roller on the back of the thigh, requesting the athlete to perform cranial and caudal movements during the established time.The intervention through the suction cups will consist of its application and produce increased flexibility of the hamstring musculature. The technique will be performed with the subject in prone position, on the stretcher, while the physiotherapist will be placed next to the member to be treated. The suckers are placed in the proximal part where the posterior musculature of the leg originates and in the distal part of the biceps femoris, semitendinosus and semimembranous insertion. This administration of the suckers will be applied during a period of 7 minutes in each member.
  Interventions: Other: Suction cups
- Foam roller (Active Comparator): The intervention will be carried out before starting the training session. The technique will be performed with the subject sitting on the floor, placing the Foam roller on the back of the thigh, requesting the athlete to perform cranial and caudal movements during the established time. The stretching exercise with the Foam roller will be done during 2 minutes in each member.
  Interventions: Other: Foam roller

INTERVENTIONS:
Other: Suction cups — The technique will be performed with the subject sitting on the floor, placing the Foam roller on the back of the thigh, requesting the athlete to perform cranial and caudal movements during the established time. The stretching exercise with the Foam roller will be done during 2 minutes in each member. The intervention through the suction cups will be performed with the subject in prone position, on the stretcher. The suckers are placed in the proximal part where the posterior musculature of the leg originates and in the distal part of the biceps femoris, semitendinosus and semimembranous insertion. This administration of the suckers will be applied during a period of 7 minutes in each member.
  Other Names: Hamstring flexibility
  Arms: Suction cups
Other: Foam roller — Each session will last 18 minutes, taking place two days a week, in a period of 4 weeks. The intervention will be carried out before starting the training session. The intervention through the self-administration of Foam roller has the objective of increasing the flexibility of the isquitibial musculature. The technique will be performed with the subject sitting on the floor, placing the Foam roller on the back of the thigh, requesting the athlete to perform cranial and caudal movements during the established time. The stretching exercise with the Foam roller will be done during 2 minutes in each member.
  Other Names: Hamstring flexibility
  Arms: Foam roller

SUMMARY:
Introduction. Basketball is a predominantly anaerobic exercise that exposes to high intensity actions (jumps, speed control, accelerations and decelerations, and changes of direction). A lack of flexibility can affect the appearance of muscle injuries. Foam roller is a myofascial self-release technique using a foam roller. The suction cups are an instrumental technique where the negative pressure produces an increase in the blood flow of the tissues.

Goals. To evaluate the effectiveness of a physiotherapy intervention through suction cups and foam roller in amateur basketball players.

Study design. Randomized, single-blind clinical study with a follow-up period. Methodology. The 20 basketball players that are expected to be recruited will be randomly assigned to the two study groups: experimental (suction cups and Foam roller) and control (Foam roller). The intervention will last 4 weeks, with 2 weekly sessions. The study variable will be: hamstring flexibility (measured with finger-ground, Well and Shober tests). The analysis of normality will be carried out with the Shapiro-Wilk test. In case of homogeneity of the groups, we will use parametric tests: t-student test of repeated measures (difference between evaluations) and ANOVA of repeated means (intra and intersubject effect).

Expected results. An intervention using suction cups and foam roller is effective in improving the flexibility of the hamstring muscles in basketball players.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 25 years
* Amateur basketball players
* Belong to the Celeste club
* Not having any injury to the hamstring musculature at the time of the study

Exclusion Criteria:

* At the time of the study they are included in a program of individualized strength training in lower limbs
* Subjects with alterations in venous return or congenital coagulopathies
* Subjects who present hypermobility
* Not signed the informed consent document

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline elongation capacity of the hamstring musculature after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The assessment of the elongation capacity of the hamstring musculature will be carried out by applying the Wells drawer or test. The subject will sit on the floor in front of the drawer, with the feet together and the plants resting on the front of the drawer, and the knees extended. Next, the athlete must tilt the trunk forward and extend the arms, sliding with outstretched hands until reaching the maximum stretch that allows its trunk flexion. The result that will be recorded corresponds to the point you can touch with your fingers. The unit of measurement for this test is the centimeter (the longer the length, the greater the hamstring elongation capacity).

SECONDARY OUTCOMES:
Change from baseline ischithiobial extensibility after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The assessment of the ischithiobial extensibility will be made by applying the finger-floor test. The subject will have to reach the greatest possible distance from the standing position with the knees in extension, by bringing the hands (by flexing the spine) towards the ground. The evaluator will measure the distance between the tip of the third finger and the floor, with the unit of measure being the centimeter (a longer length will indicate greater hamstring extensibility).
Change from baseline flexibility after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The assessment of flexibility will be measured using the Schober test. The physiotherapist will stand behind the athlete, while the subject is standing with legs extended. The evaluator will mark a line that will connect both posterior superior iliac spines, at the level of the spinous process of the fifth lumbar vertebra. Later a second mark will be made 10 centimeters away in the cranial direction to the first. Next, the subject will be asked to perform maximum flexion of the spine keeping the knees extended. When the subject is in that position of maximum column flexion, a measurement of the distance between the two marks will be made, comparing this result with the initial distance of 10 centimeters. The centimeter is the unit of measurement and a higher score indicates greater muscle flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain